CLINICAL TRIAL: NCT03591874
Title: A Phase 3 Randomized, Placebo-Controlled, Double-Masked, Multicenter, Safety and Efficacy Study of Brimonidine Tartrate Nanoemulsion Eye Drops in Patients With Ocular Graft-vs-Host Disease
Brief Title: Study of Brimonidine Tartrate Nanoemulsion Eye Drops in Patients With Ocular Graft-vs-Host Disease
Acronym: oGVHD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Primary endpoint was not met.
Sponsor: Ocugen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OCU-300-301
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Results first posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Graft Versus Host Disease; Ocular Surface Disease; oGVHD; Ocular Graft vs Host Disease; Brimonidine Tartrate; Lubricant Eye Drops; Ophthalmic Solutions; Graft vs Host Disease
Keywords: ogvhd; ocular graft vs host; Ocular Surface Disease; Ocular Graft vs Host Disease; Brimonidine Tartrate; Lubricant Eye Drops; Ophthalmic Solutions; Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Brimonidine Tartrate

STUDY DESIGN:
Intervention Model Description: This will be a randomized, placebo-controlled, double-masked, multicenter phase 3 study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects, investigators, and study personnel involved in the conduct of the study, including data management and statistics, will be masked to treatment assignment except for a specified staff member from the designated packaging vendor who will do the package labeling.
  Unmasking will be permitted in a medical emergency that requires immediate knowledge of the subject's treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OCU-300 (Experimental): Brimonidine Tartrate Nanoemulsion Eye Drops 0.18% given 2 times a day for 12 weeks.
  Interventions: Drug: Brimonidine Tartrate
- Placebos (Placebo Comparator): Placebo - Ophthalmic buffered saline Eye Drops given 2 times a day for 12 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Brimonidine Tartrate — Brimonidine Tartrate Nanoemulsion Eye Drops given 2 times a day for 12 weeks.
  Other Names: OCU-300
  Arms: OCU-300
Drug: Placebos — Opthalmic buffered saline solution Eye Drops given 2 times a day for 12 weeks.
  Other Names: Placebo (For Brimonidine Tartrate)
  Arms: Placebos

SUMMARY:
This study evaluates the use of Brimonidine tartrate nanoemulsion eye drop solution in the treatment of ocular Graft Verses Host Disease (oGVHD). Two thirds of participants will receive Brimonidine and one third will receive ophthalmic buffered saline (placebo).

DETAILED DESCRIPTION:
Ocular GVHD (oGVHD) is a common complication that occurs in 40-60% of patients who have undergone allogeneic bone marrow transplants. Driven by inflammation, oGVHD can result in damage to the ocular surface and tear-producing glands, which over time significantly diminishes quality of life and restricts daily activities due to visual impairment.

Early studies in animals and humans indicate that Brimonidine nano-emulsion, also known as OCU300, may relieve the signs and symptoms of oGVHD. These symptoms include blurry vision, foreign body sensation, burning sensation, severe light sensitivity, chronic conjunctivitis (pink or red eye), dry eyes and eye pain.

This study will be a randomized, placebo-controlled, double-masked, multicenter phase 3 study in the United States conducted at approximately 15 centers. Upon meeting the eligibility criteria, enrolled subjects with a diagnosis of definite oGVHD will be randomly assigned in a 2:1 (test: control) fashion to receive either Brimonidine Nanoemulsion Eye Drops 0.18% investigational product (test) or ophthalmic buffered saline (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years of age
* Diagnosis of definite oGVHD using the International Chronic Ocular GVHD Consensus Group Revised Diagnostic criteria in at least one eye.
* Ocular Discomfort score ≥ 3
* Validated Bulbar Redness score ≥ 40 in both eyes
* Subjects who are capable and willing to provide informed consent and follow study instructions
* Intraocular pressure (IOP) ≥ 5 mmHg and ≤22 mmHg in each eye
* Women who are not pregnant or lactating or post-menopausal or have undergone a sterilization procedure

Exclusion Criteria:

* Allergic to brimonidine or any similar products, or excipients of brimonidine
* Currently receiving any brimonidine or other treatment for glaucoma
* Receiving or have received any investigational drug or device within 30 days of screening
* Current use of contact lenses 14 days prior to screening
* Active ocular infection or ocular allergies
* Any history of eyelid surgery or ocular surgery within the past 3 months
* Corneal epithelial defect larger than 1 mm (squared) in either eye
* Received corticosteroid-containing eye drops within 14 days prior to screening or planned use during the study
* Any change in corticosteroid-containing eye drops, systemic corticosteroids/immunosuppressives, topical ocular antibiotics, cyclosporine ophthalmic emulsion 0.05% (Restasis®), cyclosporine ophthalmic solution 0.09% (Cequa®) or lifitegrast ophthalmic solution 5% (Xiidra®), or autologous serum tears within 30 days prior to screening or planned change during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-12-23 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Mayo Clinic, Phoenix, Arizona
  - Byers Eye Institute at Stanford University, Palo Alto, California
  - Emory Eye Center, Atlanta, Georgia
  - University of Kansas Medical Center, Prairie Village, Kansas
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - OHSU Casey Eye Institute | Cornea Division, Portland, Oregon
  - University of Penn Scheie Eye Institute,, Philadelphia, Pennsylvania
  - Univeristy of Pittsburgh Medical Center Eye Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Wisconsin Dept. of Ophthalmology and Visual Sciences, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
There is no current plan to share participant data with other researchers.
Supporting Information: CSR
Time Frame: A clinical Study Report will be submitted once the study data has been analyzed.

RESULTS

PARTICIPANT FLOW:
Groups:
- OCU-300: One drop of Brimonidine Tartrate Nanoemulsion 0.18% administered in each eye, two times per day (BID)
- Placebo: One drop of ophthalmic buffered saline administered in each eye BID
Period: Overall Study
Arm/Group | OCU-300 | Placebo
Started | 40 | 19
Received at Least 1 Study Treatment | 29 | 16
Completed | 21 | 12
Not Completed | 19 | 7
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Investigator Withdrawal of Subject | 1 | 0
Not completed — On Study at Time of Study Termination | 12 | 6

BASELINE CHARACTERISTICS:
Population: The safety set includes all participants who signed informed consent forms, were randomized into the study, and took at least one dose of study drug.
Groups:
- OCU-300: One drop of Brimonidine Tartrate Nanoemulsion 0.18% administered in each eye BID
- Total: Total of all reporting groups
Arm/Group | OCU-300 | Placebo | Total
Number analyzed (Participants) | 29 | 16 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (13.91) | 62.4 (7.74) | 57.3 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 21 | 10 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 16 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 28 | 15 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 84 in Validated Bulbar Redness (VBR) Score
Description: The VBR consists of a set of ten images illustrating different degrees of ocular redness, ranging from normal to severe, and each image is assigned a value from 10 (least redness) to 100 (most redness). The bulbar conjunctival injection of the participant's eye (nasal and temporal) was examined via slit-lamp examination and compared to the reference images in the VBR and graded accordingly.
Time Frame: Baseline, Day 84
Population: The Intention-To-Treat (ITT) set included all randomized participants. Here, the overall number of participants analyzed are those evaluable for this Outcome Measure and the Number Analyzed per Row is the number of participants with evaluable data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OCU-300 | Placebo
Number analyzed (Participants) | 28 | 13
score on a scale
  Baseline | 52.23 (9.238) | 51.92 (11.821)
  Day 84: number analyzed (Participants) | 21 | 12
  Day 84 | 34.88 (14.652) | 37.71 (19.378)
  Change from Baseline to Day 84: number analyzed (Participants) | 21 | 12
  Change from Baseline to Day 84 | -17.62 (14.086) | -13.96 (14.161)

2. Primary Outcome: Change From Baseline to Day 84 in Ocular Discomfort Visual Analog Scale (VAS) Score
Description: Participants were asked to rate their worst ocular pain/discomfort in the preceding 24 hours using a 10-point scale ranging from "None" (score=0) to "Unbearable/Excruciating" (score=10).
Time Frame: Baseline, Day 84
Population: The ITT set included all randomized participants. Here, the overall number of participants analyzed are those evaluable for this Outcome Measure and the Number Analyzed per Row is the number of participants with evaluable data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OCU-300 | Placebo
Number analyzed (Participants) | 28 | 13
score on a scale
  Baseline | 6.2 (1.77) | 6.5 (1.85)
  Day 84: number analyzed (Participants) | 21 | 11
  Day 84 | 4.8 (2.86) | 4.1 (3.67)
  Change from Baseline to Day 84: number analyzed (Participants) | 21 | 11
  Change from Baseline to Day 84 | -1.8 (3.33) | -2.6 (2.69)

3. Secondary Outcome: Change From Baseline to Day 84 in Symptom Assessment iN Dry Eye (SANDE) Questionnaire Scores
Description: The SANDE questionnaire is a short VAS assessment that quantifies both severity and frequency of current dry eye symptoms. The SANDE is comprised of two questions, and each question employs a 100-mm horizontal linear VAS. The measurement of symptom frequency ranges from "rarely" to "all of the time", and the symptom severity from "very mild" to "very severe". Data collected from the SANDE questionnaire was calculated by multiplying the frequency score by the severity score and obtaining the square root. The result is the Overall SANDE score which ranges from 0 to 100, with 100 being the maximal amount of dry eye symptoms and 0 being the minimal amount of dry eye symptoms.
Time Frame: Baseline, Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OCU-300 | Placebo
Number analyzed (Participants) | 28 | 13
score on a scale
  Baseline | 74.4 (18.97) | 69.1 (21.90)
  Day 84: number analyzed (Participants) | 19 | 10
  Day 84 | 50.5 (24.05) | 44.1 (36.43)
  Change from Baseline to Day 84: number analyzed (Participants) | 19 | 10
  Change from Baseline to Day 84 | -26.5 (22.24) | -26.6 (27.50)

ADVERSE EVENTS:
Time Frame: Day 1 (post-dose) up to 84 Days
Arm/Group | OCU-300 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/29 | 1/16
Other Adverse Events (participants affected / at risk) | 1/29 | 4/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OCU-300 (N=29) | Placebo (N=16)
Gastrointestinal infection (Infections and infestations) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OCU-300 (N=29) | Placebo (N=16)
Influenza (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT03591874/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT03591874/SAP_001.pdf